CLINICAL TRIAL: NCT01593449
Title: A Community-based Social Networking Intervention to Increase Walking in Dog Owners
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Massachusetts, Lowell (Other)
Responsible Party: Principal Investigator, Kristin Schneider, Principal Investigator, Rosalind Franklin University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIH 5 UL1RR031982-02
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Sedentary
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- American Heart Association (Active Comparator): Participants will receive handouts on increasing physical activity derived from the American Heart Association materials on increasing physical activity.
  Interventions: Behavioral: Community-based social networking intervention
- Dog Walking (Experimental): The 6-month dog walking intervention involves 5 components to address the individual, interpersonal and community levels of the socio-ecological model: newsletters, pedometers, social networking website, neighborhood dog walks, and invitations to community events.
  Interventions: Behavioral: Community-based social networking intervention

INTERVENTIONS:
Behavioral: Community-based social networking intervention — Participation in this study lasts for 7 months and includes a baseline visit, an orientation visit, the 6 month intervention, and a 6 month assessment visit.

SUMMARY:
The present study aims to initially test a community dog walking intervention that addresses individual, interpersonal and community factors associated with dog walking. The study will be conducted in two cities, Worcester and Lowell, as a collaboration between investigators from UMass Medical School and UMass-Lowell.

DETAILED DESCRIPTION:
This is a group randomized trial where 8 communities in Worcester and Lowell (4 per city) will be randomly assigned to the 6-month dog walking intervention or a standard, self-help, print-based physical activity control condition. Dog owners (N=120; 15 per community) will be recruited. The intervention includes a social networking website, monthly newsletters, twice monthly neighborhood dog walks and community events. The intervention will: 1) educate owners about the benefits of dog walking to themselves and their dog, 2) teach strategies for regular dog walking, 3) teach dog walking tips and provide dog training seminars, 4) promote self-monitoring and goal setting for dog walking, 5) provide social networking opportunities for dog owners and 6) promote a sense of community via participation in neighborhood dog walks and community events. Intervention feasibility will be assessed by measures of implementation success, including recruitment and retention rates, website use, intervention satisfaction and attendance at neighborhood walks and community events. Initial efficacy will be assessed via change in weekly steps measured via a pedometer from baseline to 6-months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will own a dog that is in good health and considered a household pet, be a Worcester or Lowell resident, be aged > 21 years old and have home internet access. Participants with cardiovascular disease, diabetes or other chronic health condition are eligible with permission from their PCP to participate.

Exclusion Criteria:

Participants will be excluded for any of the following:

1. Inability or unwillingness to give informed consent
2. Plans to move out of the area within the study period
3. Participated in a focus group during the developmental phase
4. Another household member is participating in the study
5. Pregnant or planning a pregnancy in the next six months
6. Condition that inhibits exercise (e.g., unable to walk unaided, or cannot walk 1/4 mile without stopping)
7. Incapable of engaging in physical activity as assessed by the Physical Activity Readiness Questionnaire
8. Self-report engaging in > 150 minutes of moderate and vigorous intensity physical activity per week.
9. The participant's dog has a history of biting a human or has not received a rabies vaccination.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
feasibility | 6 months
  Feasibility will be assessed by implementation success, including recruitment and retention rates, website use, intervention satisfaction and attendance at neighborhood walks and community events.

SECONDARY OUTCOMES:
Weekly steps | baseline and 6 months
  Pedometers that record 7-days of data will be used to measure steps at baseline and 6 months
weekly dog walking minutes | baseline and 6 months
  Self-reported minutes of dog walking measured using the DAPA tool.
social support for walking | baseline and 6 months
  Self-reported social support for walking
sense of community | baseline and 6 months
  self-reported sense of community

CONTACTS AND LOCATIONS:
Overall Officials: Krisitin Schneider, Ph.D., Principal Investigator — Rosalind Franklin Medical School
Locations (2):
- United States (2):
  - University of Massachusetts Lowell, Lowell, Massachusetts
  - University of Massachusetts Medical Schol, Worcester, Massachusetts

REFERENCES:
- [Derived] Schneider KL, Murphy D, Ferrara C, Oleski J, Panza E, Savage C, Gada K, Bozzella B, Olendzki E, Kern D, Lemon SC. An online social network to increase walking in dog owners: a randomized trial. Med Sci Sports Exerc. 2015 Mar;47(3):631-9. doi: 10.1249/MSS.0000000000000441. PMID 25003777